CLINICAL TRIAL: NCT04873258
Title: Development of a Non-invasive Screening Tool to Predict Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD) in Volunteers on Clinical Trials Utilising Machine-learning and Bioimpedance Vector Analysis
Brief Title: Development of a Non-invasive Screening Tool to Predict Metabolic Dysfunction-associated Steatotic Liver Disease
Acronym: MASLD
Status: Recruiting | Type: Observational
Sponsor: Richmond Research Institute (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Organization: Richmond Pharmacology Limited (Industry)
Other Study IDs: C19030
Record Dates: First submitted 2021-04-20; First posted 2021-05-05 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Fatty Liver; MASLD; MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Obesity and Obesity-related Medical Conditions
Keywords: Fatty liver; MASLD
MeSH Terms: conditions — Fatty Liver; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with MASLD: Patients with known MASLD
  Interventions: Diagnostic Test: Bioimpedence Vector Analysis
- Healthy volunteers: Patients without any known health issues
  Interventions: Diagnostic Test: Bioimpedence Vector Analysis

INTERVENTIONS:
Diagnostic Test: Bioimpedence Vector Analysis — Bioimpedence vector analysis

SUMMARY:
A generic screening study to establish structural and/or functional baselines of specific organs.

DETAILED DESCRIPTION:
Fatty liver disease is a common condition (25% of the population) which can lead to liver inflammation, liver scarring and even liver cancer. Clinical trials are often performed in healthy volunteers, who may have underlying fatty liver without knowledge of it. In clinical trials fatty liver can both mean volunteers have abnormal liver tests, preventing them joining the trial, as well as more likely to have a possible liver drug reaction, causing volunteers to withdraw from a clinical trial of a new drug.

The principal objective of the study is to develop a clinical scoring tool that can accurately predict fatty liver disease in study volunteers, without the need for invasive tests (such as a tissue biopsy).

We aim to recruit initially 2000 volunteers to this study, both healthy volunteers and patients with known MASLD.

Volunteers will attend the unit to undergo all assessments on one day. Once consent is given with a study research physician, bloods will be taken and body measurements made (including BMI, weight, waist circumference). A full medical history and physical examination will then be performed by the research physician.

Bioimpedance body composition analysis will then be performed on an ACUNIQ device. Finally ultrasound of the liver and fibroscan will be performed. Once all assessments are complete the study volunteer will be discharged from the unit.

Once all results are finalised, analysis will be performed on all the data to create a clinical score to predict the presence of MASLD, both with statistical and machine learning methods.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged ≥18 to ≤80 years at the date of signing the informed consent.
2. Willingness and ability to provide written, personally signed, and dated informed consent, in accordance with the latest ICH Good Clinical Practice (GCP) Guidelines and applicable regulations.
3. An understanding, ability and willingness to fully comply with project procedures and restrictions.

For PART B only:

1. With a known history of MASLD as evidenced either of:

1. GP diagnosis on HCF
2. Documented Fibroscan or liver US demonstrating MASLD

Exclusion Criteria:

1. Known alcoholic liver disease, history of cirrhosis of any other cause (metabolic, viral hepatitis or other)
2. Any other significant previous liver pathology (liver malignancy, portal hypertension, infiltrative liver disease)
3. Alcohol consumption >30 units per week
4. An Implanted cardiac devices

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult male or female volunteers for other clinical trials taking place at the study unit.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Establishment of Classification Tool for Use in Clinical Trials | Study duration (1 year)
  The success of the final classification tool (as measured by area under the receiver operator curve (AUROC). The initial measure to generate the dataset will be the presence or absence of MASLD on liver USS.

SECONDARY OUTCOMES:
Normal LFT Range in NAFLD patients | Study duration (1 year)
  The normal range of LFT's in patients with known NAFLD

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Taubel, MD, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd. 1a Newcomen St, London Bridge, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No